CLINICAL TRIAL: NCT01793610
Title: A Randomized, Double-Blind, Dose Response Phase 2 Pilot Study of Manualized MDMA-Assisted Psychotherapy in Subjects With Chronic, Treatment-Resistant Posttraumatic Stress Disorder (PTSD)
Brief Title: Dose-Response Study of MDMA-assisted Psychotherapy in People With PTSD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lykos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MP-12
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Results first posted 2020-10-14 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Posttraumatic Stress Disorder
Keywords: MDMA; Posttraumatic stress disorder; sleep; Depression; Safety
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Psychotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Comparator Dose (40 mg) MDMA-assisted therapy (Active Comparator): Participants receive an initial dose of comparator dose midomafetamine HCl (40 mg) during each of two therapy sessions.
  Interventions: Drug: Comparator Dose (40mg) MDMA HCl; Behavioral: Psychotherapy
- Active Dose 2 (100 mg) MDMA-assisted therapy (Experimental): Participants receive an initial dose of Active Dose 2 midomafetamine HCl (100 mg) during each of two therapy sessions.
  Interventions: Drug: Active Dose 2 (100 mg) MDMA HCl; Behavioral: Psychotherapy
- Active Dose 1 (125 mg) MDMA-assisted therapy (Experimental): Participants receive an initial dose of Active Dose 1 midomafetamine HCl (125 mg) during each of two therapy sessions.
  Interventions: Drug: Active Dose 1 (125 mg) MDMA HCl; Behavioral: Psychotherapy

INTERVENTIONS:
Drug: Comparator Dose (40mg) MDMA HCl — An initial comparator-dose of 40 mg midomafetamine HCl orally given at the start of two separate psychotherapy sessions scheduled 3 to 5 weeks apart, with the initial dose possibly followed 1.5 to 2.5 hours later by a supplemental dose half the size of the initial dose (20 mg).
  Other Names: 3,4-methylenedioxymethamphetamine; midomafetamine HCl; midomafetamine; MDMA
  Arms: Comparator Dose (40 mg) MDMA-assisted therapy
Drug: Active Dose 2 (100 mg) MDMA HCl — An initial dose of full-dose 100 mg midomafetamine HCl orally given at the start of two separate psychotherapy sessions scheduled 3 to 5 weeks apart, with the initial dose possibly followed 1.5 to 2.5 hours later by a supplemental dose half the size of the initial dose (50 mg).
  Other Names: 3,4-methylenedioxymethamphetamine; midomafetamine HCl; midomafetamine; MDMA
  Arms: Active Dose 2 (100 mg) MDMA-assisted therapy
Drug: Active Dose 1 (125 mg) MDMA HCl — An initial dose of full-dose 125 mg midomafetamine HCl orally given at the start of two separate psychotherapy sessions scheduled 3 to 5 weeks apart, with the initial dose possibly followed 1.5 to 2.5 hours later by a supplemental dose half the size of the initial dose (62.5 mg).
  Other Names: 3,4-methylenedioxymethamphetamine; midomafetamine HCl; midomafetamine; MDMA
  Arms: Active Dose 1 (125 mg) MDMA-assisted therapy
Behavioral: Psychotherapy — Non-directive manualized therapy
  Other Names: Manualized MDMA-assisted psychotherapy

SUMMARY:
The goal of this clinical trial is to learn if MDMA in combination with therapy is safe and effective in people with chronic, treatment-resistant PTSD.

The main questions it aims to answer are:

* Does MDMA-assisted therapy reduce PTSD symptoms?
* Is there a difference in PTSD symptoms between the 40 mg, 100 mg, and 125 mg groups?

Researchers will compare two active doses (100 mg and 125 mg) of MDMA-assisted therapy versus a comparator dose of 40 mg MDMA-assisted therapy to determine if there is a reduction in PTSD symptoms.

Participants will undergo three non-drug preparatory sessions, three MDMA-assisted therapy sessions and three non-drug integrative therapy sessions after each MDMA-assisted therapy session.

DETAILED DESCRIPTION:
This Phase 2 pilot study is a randomized, double-blind, dose response study to examine the safety and efficacy of MDMA-assisted psychotherapy in 23 subjects with chronic, treatment-resistant PTSD of at least six months duration. This study assessed two active doses of MDMA, active dose 1 (100 mg) and active dose 2 (125 mg), to a comparator dose of MDMA (40 mg) during psychotherapy sessions. The initial dose of MDMA was followed 1.5 to 2.5 hours later by an optional supplemental dose of MDMA that was half the size of the first dose. MDMA was administered orally in two experimental sessions lasting up to eight hours and scheduled three to five weeks apart.

Subjects were prepared for MDMA-assisted psychotherapy in three preparatory sessions prior to the first experimental session, and worked with the same pair of therapists throughout the study. After each experimental session, three integrative sessions were scheduled with the subject, including one integrative session the morning after the experimental session. During integrative sessions, subjects processed and connected their thoughts and feelings about the experience with their therapist team.

Subjects who received the comparator dose (40 mg) were given the option to enroll in Stage 2, where they underwent three open-label MDMA-assisted psychotherapy sessions. 100 mg of MDMA was administered in the first session and therapists determined whether to increase to 125 mg of MDMA for the second and third experimental sessions. People who received 125 mg of MDMA during the first two experimental sessions received the same dose during an open-label third experimental session. People who received 100 mg of MDMA during the first two sessions were able to choose, in consultation with their therapist, to either continue to receive 100 mg in a third session or to increase their dose to 125 mg.

A blinded independent rater (IR) assessed the severity of PTSD symptoms at baseline, one month after the second experimental session (the primary endpoint), two months after the third open-label experimental session, and at equivalent points in Stage 2.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic PTSD for six months or longer.
* Have a CAPS score showing moderate to severe PTSD symptoms.
* At least one unsuccessful attempt at treatment for PTSD either with talk therapy or with drugs, or discontinuing treatment because of inability to tolerate psychotherapy or drug therapy.
* Are at least 18 years old.
* Must be generally healthy.
* Are willing to refrain from taking any psychiatric medications during the study period.
* Willing to follow restrictions and guidelines concerning consumption of food, beverages or nicotine the night before and just prior to each MDMA session.
* Willing to remain overnight at the study site.
* Are willing to be driven home after experimental sessions either by a driver they arrange, a taxi, or study personnel.
* Are willing to be contacted via telephone by study personnel.
* If of child-bearing age, must have a negative pregnancy and agree to use an effective form of birth control.
* Must provide a personal contact who is willing to be reached in case of emergency.
* Agree to let the investigators know within 48 hours of any planned medical interventions.
* Are proficient in reading and speaking English.
* Agree to have all psychotherapy sessions recorded.
* Agree not to participate in any other interventional clinical trials during the course of the study.

Exclusion Criteria:

* Are pregnant or nursing, or if of child-bearing age and do not use an effective means of birth control.
* Weigh less than 48 kg.
* Meet DSM-IV criteria for substance abuse or dependence for any substance in the past 60 days.
* Have used "Ecstasy" (material represented as containing MDMA) more than five times in the last ten years or at least once within 6 months of the MDMA session.
* Are unable to give adequate informed consent.
* Upon review of past and current drugs/medication, must not be on or have taken a medication that is exclusionary.
* Upon review of medical or psychiatric history, must not have any current or past diagnosis that would be considered a risk to participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-05-13 (Actual); Primary Completion 2015-12-03 (Actual); Study Completion 2017-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcela d'Otalora, MA, LPC, Principal Investigator — Private Practice
Locations (1):
- Offices of Marcela d'Otalora, Boulder, Colorado, United States

REFERENCES:
- [Background] Blake DD, Weathers FW, Nagy LM, Kaloupek DG, Gusman FD, Charney DS, Keane TM. The development of a Clinician-Administered PTSD Scale. J Trauma Stress. 1995 Jan;8(1):75-90. doi: 10.1007/BF02105408. PMID 7712061
- [Background] Beck AT, Steer RA. Internal consistencies of the original and revised Beck Depression Inventory. J Clin Psychol. 1984 Nov;40(6):1365-7. doi: 10.1002/1097-4679(198411)40:63.0.co;2-d. PMID 6511949
- [Background] Beck AT, Steer RA, Ball R, Ranieri W. Comparison of Beck Depression Inventories -IA and -II in psychiatric outpatients. J Pers Assess. 1996 Dec;67(3):588-97. doi: 10.1207/s15327752jpa6703_13. PMID 8991972
- [Derived] Jerome L, Feduccia AA, Wang JB, Hamilton S, Yazar-Klosinski B, Emerson A, Mithoefer MC, Doblin R. Long-term follow-up outcomes of MDMA-assisted psychotherapy for treatment of PTSD: a longitudinal pooled analysis of six phase 2 trials. Psychopharmacology (Berl). 2020 Aug;237(8):2485-2497. doi: 10.1007/s00213-020-05548-2. Epub 2020 Jun 4. PMID 32500209
- [Derived] Feduccia AA, Jerome L, Yazar-Klosinski B, Emerson A, Mithoefer MC, Doblin R. Breakthrough for Trauma Treatment: Safety and Efficacy of MDMA-Assisted Psychotherapy Compared to Paroxetine and Sertraline. Front Psychiatry. 2019 Sep 12;10:650. doi: 10.3389/fpsyt.2019.00650. eCollection 2019. PMID 31572236
- [Derived] Mithoefer MC, Feduccia AA, Jerome L, Mithoefer A, Wagner M, Walsh Z, Hamilton S, Yazar-Klosinski B, Emerson A, Doblin R. MDMA-assisted psychotherapy for treatment of PTSD: study design and rationale for phase 3 trials based on pooled analysis of six phase 2 randomized controlled trials. Psychopharmacology (Berl). 2019 Sep;236(9):2735-2745. doi: 10.1007/s00213-019-05249-5. Epub 2019 May 7. PMID 31065731

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Candidates were recruited via Internet advertisements and referrals from mental health professionals.
Groups:
- Comparator Dose MDMA (40 mg) and Psychotherapy: Participants receive an initial dose of 40 mg of MDMA orally, with an optional supplemental dose of 20 mg MDMA 1.5 to 2.5 hours later.
- Active Dose 2 MDMA (100 mg) and Psychotherapy: Participants receive an initial dose of 100 mg of MDMA orally, with an optional supplemental dose of 50 mg MDMA 1.5 to 2.5 hours later.
- Active Dose 1 MDMA (125 mg) and Psychotherapy: Participants receive an initial dose of 125 mg of MDMA orally, with an optional supplemental dose of 62.5 mg MDMA 1.5 to 2.5 hours later.
Period: Stage 1 Randomized, Double-blind Period
Arm/Group | Comparator Dose MDMA (40 mg) and Psychotherapy | Active Dose 2 MDMA (100 mg) and Psychotherapy | Active Dose 1 MDMA (125 mg) and Psychotherapy
Started | 6 | 9 | 13
Completed | 6 | 9 | 12
Not Completed | 0 | 0 | 1
Period: Stage 2 Open-Label Crossover Period
Arm/Group | Comparator Dose MDMA (40 mg) and Psychotherapy | Active Dose 2 MDMA (100 mg) and Psychotherapy | Active Dose 1 MDMA (125 mg) and Psychotherapy
Started (Only Comparator Dose participants were included in Stage 2. Stage 2 cross-over occurred approximately one month following the Stage 1 Primary Endpoint visit. One Comparator Dose participant did not participate in Stage 2.) | 5 | 0 | 0
Completed | 5 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT)
Groups:
- Comparator-dose MDMA (40 mg) and Psychotherapy: Participants receive an initial dose of 40 mg of MDMA orally, with an optional supplemental dose of 20 mg MDMA 1.5 to 2.5 hours later.
- Total: Total of all reporting groups
Arm/Group | Active Dose 1 MDMA (125 mg) and Psychotherapy | Active Dose 2 MDMA (100 mg) and Psychotherapy | Comparator-dose MDMA (40 mg) and Psychotherapy | Total
Number analyzed (Participants) | 12 | 9 | 6 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (15.53) | 39.6 (9.8) | 40 (11.71) | 42.4 (12.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 5 | 19
  Male | 4 | 3 | 1 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 12 | 8 | 6 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 11 | 9 | 5 | 25
  American Indian Or Alaska Native | 0 | 0 | 1 | 1
  Other | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinician Administered PTSD Scale for DSM-IV (CAPS-IV) Total Severity Score From Baseline to One Month Post 2nd Experimental Session
Description: The Clinician-Administered PTSD Scale for DSM-IV (CAPS-IV) is a clinician administered and scored assessment of PTSD symptoms via structured interview based upon PTSD diagnosis in DSM-IV. It contains symptom subscales, a CAPS-IV total severity score, and a diagnostic score. The total severity score is a sum of symptom frequency and intensity scores for the subscales B (re-experiencing), C (avoidance) and D (hypervigilance) and ranges from 0 to 136, with higher scores indicating greater severity of PTSD symptoms.
Time Frame: Baseline Enrollment to 1-Month Post 2nd Experimental Session (Stage 1 Primary Endpoint)
Population: Modified Intent-to-Treat set (mITT), Stage 1 participants
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Active Dose 1 (125 mg) MDMA and Psychotherapy: Participants receive an initial dose of 125 mg of MDMA orally, with an optional supplemental dose of 62.5 mg MDMA 1.5 to 2.5 hours later.
- Active Dose 2 (100 mg) MDMA and Psychotherapy: Participants receive an initial dose of 100 mg of MDMA orally, with an optional supplemental dose of 50 mg MDMA 1.5 to 2.5 hours later.
- Comparator-dose (40 mg) MDMA and Psychotherapy: Participants receive an initial dose of 40 mg of MDMA orally, with an optional supplemental dose of 20 mg MDMA 1.5 to 2.5 hours later.
Arm/Group | Active Dose 1 (125 mg) MDMA and Psychotherapy | Active Dose 2 (100 mg) MDMA and Psychotherapy | Comparator-dose (40 mg) MDMA and Psychotherapy
Number analyzed (Participants) | 12 | 9 | 6
score on a scale | -26.3 (29.52) | -24.4 (24.22) | -11.5 (21.21)

2. Secondary Outcome: Change in PTSD Diagnostic Scale (PDS) From Baseline to One Month Post 2nd Experimental Session
Description: The PTSD Diagnostic Scale (PSD) is self-report measure designed to follow DSM-IV criteria for assessing PTSD. It contains 49 items, with responses made on a four-point scale, ranging from 0 ("not at all") to 3 ("five or more times a week"). The PDS consists of a list of 12 potential traumatic events, 12 items addressing elements of the traumatic event, 17 symptom items, and 9 items assessing impact on areas of life function. Items addressing elements of the traumatic event and life function are answered as either present or not present (Yes or No). The 17 items are summed to create a symptom severity score, with higher scores indicating a greater number and/or intensity of PTSD symptoms. The symptom severity score ranges from 0 to 51.
Time Frame: Baseline Enrollment to 1-Month Post 2nd Experimental Session (Stage 1 Primary Endpoint)
Population: Modified Intent-to-Treat set (mITT), Stage 1 participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Dose 1 (125 mg) MDMA and Psychotherapy | Active Dose 2 (100 mg) MDMA and Psychotherapy | Comparator-dose (40 mg) MDMA and Psychotherapy
Number analyzed (Participants) | 12 | 9 | 6
score on a scale | -11.3 (11.26) | -10.0 (10.44) | -4.2 (3.13)

3. Secondary Outcome: Change in Beck Depression Inventory II (BDI-II) From Baseline to One Month Post 2nd Experimental Session
Description: Validated self-report measure of symptoms of depression. The BDI-II total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe depressive symptoms. The scores range from 0 to 63, with higher score indicating greater severity of depressive symptoms.
Time Frame: Baseline Enrollment to 1-Month Post 2nd Experimental Session (Stage 1 Primary Endpoint)
Population: Modified Intent-to-Treat set (mITT), Stage 1 participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Dose 1 (125 mg) MDMA and Psychotherapy | Active Dose 2 (100 mg) MDMA and Psychotherapy | Comparator-dose (40 mg) MDMA and Psychotherapy
Number analyzed (Participants) | 12 | 9 | 6
score on a scale | -11.0 (13.68) | -9.9 (13.26) | -11.5 (7.79)

4. Secondary Outcome: Change in Global Assessment of Functioning (GAF) Total Score From Baseline to One Month Post 2nd Experimental Session
Description: The Global Assessment of Functioning (GAF) Scale is a numeric scale ranging from 0 through 100 that is used by mental health clinicians and physicians to subjectively rate the social, occupational, and psychological functioning of adults. Higher scores indicate better functioning.
Time Frame: Baseline Enrollment to 1-Month Post 2nd Experimental Session (Stage 1 Primary Endpoint)
Population: Modified Intent-to-Treat set (mITT), Stage 1 participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Dose 1 (125 mg) MDMA-assisted Therapy | Active Dose 2 (100 mg) MDMA-assisted Therapy | Comparator Dose (40 mg) MDMA-assisted Therapy
Number analyzed (Participants) | 12 | 9 | 6
score on a scale | 0.6 (10.57) | 2.4 (9.63) | 1.5 (4.59)

5. Secondary Outcome: Change in Pittsburgh Sleep Quality Index (PSQI) From Baseline to One Month Post 2nd Experimental Session
Description: The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances. It is comprised of 18 items that yield seven component scores. Component scores are summed to create a total score. Total scores range from 0 (better) to 21 (worse), with higher scores indicating poor sleep quality.
Time Frame: Baseline Enrollment to 1-Month Post 2nd Experimental Session (Stage 1 Primary Endpoint)
Population: Modified Intent-to-Treat set (mITT), Stage 1 participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Dose 1 (125 mg) MDMA and Psychotherapy | Active Dose 2 (100 mg) MDMA and Psychotherapy | Comparator-dose (40 mg) MDMA and Psychotherapy
Number analyzed (Participants) | 12 | 9 | 6
score on a scale | -2.0 (4.69) | -3.6 (6.19) | -0.8 (2.48)

6. Secondary Outcome: Change in Dissociative Experiences Scale (DES-II) From Baseline to One Month Post 2nd Experimental Session
Description: The DES-II is a 28-item self-report measure of dissociation, defined as a lack of normal integration of an individual's thoughts, feelings, or experiences into the stream of consciousness or memory. The scale consists of statements describing facets of dissociation. Respondents indicate how often the specific experience happens to them, from "never" to "always." The DES-II uses the same items but with responses made on a 10 point scale from "0%" to "100%" of the time. The scale is scored by treating percentages as single digits to produce a total score with higher scores indicating greater severity. The total score ranges from 0 to 100.
Time Frame: Baseline Enrollment to 1-Month Post 2nd Experimental Session (Stage 1 Primary Endpoint)
Population: Modified Intent-to-Treat set (mITT), Stage 1 participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Dose 1 (125 mg) MDMA-assisted Therapy | Active Dose 2 (100 mg) MDMA-assisted Therapy | Comparator Dose (40 mg) MDMA-assisted Therapy
Number analyzed (Participants) | 12 | 9 | 6
score on a scale | -5.9 (11.98) | -13.3 (15.25) | -0.2 (6.95)

7. Secondary Outcome: Change in Posttraumatic Growth Inventory (PTGI) From Baseline to One Month Post 2nd Experimental Session
Description: The PTGI is a 21-item self-report measure of perceived growth or benefits occurring after a traumatic event. It contains five subscales: relationship to others, new possibilities, personal strength, spiritual change, and appreciation of life. PTGI scores on a 6 point scale are: 0 - I did not experience this as a result of my crisis; 1 - I experienced this change to a very small degree as a result of my crisis; 2 - I experienced this change to a small degree as a result of my crisis; 3 - I experienced this change to a moderate degree as a result of my crisis; 4 - I experienced this change to a great degree as a result of my crisis; and 5 - I experienced this change to a very great degree as a result of my crisis. A total score is calculated by summing the responses to all 21 items, each rated on a 6-point scale, with higher scores indicating greater post-traumatic growth
Time Frame: Baseline Enrollment to 1-Month Post 2nd Experimental Session (Stage 1 Primary Endpoint)
Population: Modified Intent-to-Treat set (mITT), Stage 1 participants. 1 Comparator Dose participant did not complete a baseline PTGI assessment so is excluded from this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Dose 1 (125 mg) MDMA-assisted Therapy | Active Dose 2 (100 mg) MDMA-assisted Therapy | Comparator Dose (40 mg) MDMA-assisted Therapy
Number analyzed (Participants) | 10 | 9 | 5
score on a scale | 15.0 (19.71) | 16.2 (29.47) | 3.8 (24.65)

ADVERSE EVENTS:
Time Frame: All AEs from baseline to long-term follow-up (approximately 18 months)
Groups:
- Active Dose 1 MDMA (125 mg) and Psychotherapy (Stage 1): Participants receive an initial dose of 125 mg of midomafetamine HCl orally, with an optional supplemental dose of 62.5 mg 1.5 to 2.5 hours later during two blinded sessions.
- Active Dose 2 MDMA (100 mg) and Psychotherapy (Stage 1): Participants receive an initial dose of 100 mg of midomafetamine HCl orally, with an optional supplemental dose of 50 mg 1.5 to 2.5 hours later during two blinded sessions.
- Comparator-dose MDMA (40 mg) and Psychotherapy (Stage 1): Participants receive an initial dose of 40 mg of midomafetamine HCl orally, with an optional supplemental dose of 20 mg 1.5 to 2.5 hours later during two blinded sessions.
- Open-Label Session: Active Dose 1: Participants will receive one open-label MDMA-assisted therapy session with an initial dose of 125 mg of midomafetamine HCl orally, with an optional supplemental dose of 62.5 mg 1.5 to 2.5 hours later.
- Open-Label Session: Active Dose 2: Participants will receive one open-label MDMA-assisted therapy session with an initial dose of 100 mg of midomafetamine HCl orally, with an optional supplemental dose of 62.5 mg 1.5 to 2.5 hours later.
- Crossover Open-Label Sessions: Comparator Dose: Participants who received the comparator dose during Stage 1 will have the opportunity to crossover and take part in a second study segment, referred to as Stage 2, with three open-label MDMA-assisted therapy sessions.
  In the first session, the dose will be 100 mg followed 1.5 to 2.5 hours later by an optional supplement dose of 50 mg.
  In the second and third sessions, participants will have the option to keep the same dose or titrate up to 125 mg, followed 1.5 to 2.5 hours later by 62.5 mg.
- 12 Month Follow-up: Active Dose 1; 12 Month Follow-up: Active Dose 2: Adverse events collected 12 months after the participant's final MDMA-assisted therapy session.
- 12 Month Follow-up: Comparator Dose: Adverse events collected 12 months after the participant's final MDMA-assisted therapy session (following crossover to receive 3 additional treatment sessions with active dose).
- SRRs: Active Dose 1; SRRs: Active Dose 2; SRRs: Comparator: Spontaneously reported reactions (SRRs) on open-label experimental sessions days and 7 days after.
Arm/Group | Active Dose 1 MDMA (125 mg) and Psychotherapy (Stage 1) | Active Dose 2 MDMA (100 mg) and Psychotherapy (Stage 1) | Comparator-dose MDMA (40 mg) and Psychotherapy (Stage 1) | Open-Label Session: Active Dose 1 | Open-Label Session: Active Dose 2 | Crossover Open-Label Sessions: Comparator Dose | 12 Month Follow-up: Active Dose 1 | 12 Month Follow-up: Active Dose 2 | 12 Month Follow-up: Comparator Dose | SRRs: Active Dose 1 | SRRs: Active Dose 2 | SRRs: Comparator
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/9 | 0/6 | 0/12 | 0/9 | 0/5 | 0/11 | 0/9 | 0/5 | 0/13 | 0/9 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/9 | 0/6 | 0/12 | 1/9 | 0/5 | 0/11 | 1/9 | 0/5 | 0/13 | 0/9 | 0/6
Other Adverse Events (participants affected / at risk) | 8/13 | 6/9 | 1/6 | 5/12 | 3/9 | 3/5 | 2/11 | 1/9 | 1/5 | 0/13 | 0/9 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Dose 1 MDMA (125 mg) and Psychotherapy (Stage 1) (N=13) | Active Dose 2 MDMA (100 mg) and Psychotherapy (Stage 1) (N=9) | Comparator-dose MDMA (40 mg) and Psychotherapy (Stage 1) (N=6) | Open-Label Session: Active Dose 1 (N=12) | Open-Label Session: Active Dose 2 (N=9) | Crossover Open-Label Sessions: Comparator Dose (N=5) | 12 Month Follow-up: Active Dose 1 (N=11) | 12 Month Follow-up: Active Dose 2 (N=9) | 12 Month Follow-up: Comparator Dose (N=5) | SRRs: Active Dose 1 (N=13) | SRRs: Active Dose 2 (N=9) | SRRs: Comparator (N=6)
Ruptured ovarian cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Active Dose 1 MDMA (125 mg) and Psychotherapy (Stage 1) (N=13) | Active Dose 2 MDMA (100 mg) and Psychotherapy (Stage 1) (N=9) | Comparator-dose MDMA (40 mg) and Psychotherapy (Stage 1) (N=6) | Open-Label Session: Active Dose 1 (N=12) | Open-Label Session: Active Dose 2 (N=9) | Crossover Open-Label Sessions: Comparator Dose (N=5) | 12 Month Follow-up: Active Dose 1 (N=11) | 12 Month Follow-up: Active Dose 2 (N=9) | 12 Month Follow-up: Comparator Dose (N=5) | SRRs: Active Dose 1 (N=13) | SRRs: Active Dose 2 (N=9) | SRRs: Comparator (N=6)
Anxiety (Psychiatric disorders) | 3 | 3 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0/12 | 0 | 5/5
Headache (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0/12 | 0 | 2/5
Nausea (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0/12 | 0 | 0/5
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incorrect dose administered (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Obsessive rumination (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0/12 | 0 | 1/5
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeling abnormal (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post concussion syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Difficulty Concentrating (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0/12 | 0 | 2/5
Drowsiness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0/12 | 0 | 1/5
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0/12 | 0 | 2/5
Impaired Judgment (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0/12 | 0 | 1/5
Insomnia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0/12 | 0 | 3/5
Jaw Clenching, Tight Jaw (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0/12 | 0 | 2/5
Lack of Appetite (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0/12 | 0 | 1/5
Low mood (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0/12 | 0 | 2/5
Muscle tension (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0/12 | 0 | 1/5
Need more sleep (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0/12 | 0 | 2/5
Perspiration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0/12 | 0 | 1/5
Ruminations (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0/12 | 0 | 2/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2014-08-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT01793610/Prot_003.pdf
  • Statistical Analysis Plan (2016-02-26): https://cdn.clinicaltrials.gov/large-docs/10/NCT01793610/SAP_000.pdf
  • Informed Consent Form (2016-07-18): https://cdn.clinicaltrials.gov/large-docs/10/NCT01793610/ICF_004.pdf